CLINICAL TRIAL: NCT04862663
Title: A Phase Ib/III, Open-label, Randomised Study of Capivasertib Plus CDK4/6 Inhibitors and Fulvestrant Versus CDK4/6 Inhibitors and Fulvestrant in Hormone Receptor-Positive and Human Epidermal Growth Factor Receptor 2-Negative Locally Advanced, Unresectable or Metastatic Breast Cancer (CAPItello-292)
Brief Title: Capivasertib + CDK4/6i + Fulvestrant for Advanced/Metastatic HR+/HER2- Breast Cancer (CAPItello-292)
Acronym: CAPItello-292
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D361DC00001; 2020-004637-20 (EudraCT Number)
Record Dates: First submitted 2021-03-17; First posted 2021-04-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced (Inoperable) or Metastatic Breast Cancer
Keywords: Locally advanced (inoperable) or Metastatic Breast Cancer
MeSH Terms: interventions — capivasertib; Fulvestrant; palbociclib; ribociclib; abemaciclib

STUDY DESIGN:
Intervention Model Description: Phase Ib: Open, Parallel groups allowed, recruiting up to approx. 222 participants.
  Phase III: open-label, randomised, recruiting approx. 794 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Capivasertib Plus Palbociclib and Fulvestrant (Experimental): Capivasertib Plus Palbociclib and Fulvestrant (Ph 1b)
  Interventions: Drug: Capivasertib; Drug: Fulvestrant; Drug: Palbociclib
- Capivasertib Plus Ribociclib and Fulvestrant (Experimental): Capivasertib Plus Ribociclib and Fulvestrant (Ph 1b)
  Interventions: Drug: Ribociclib
- Capivasertib Plus Abemaciclib and Fulvestrant (Experimental): Capivasertib Plus Abemaciclib and Fulvestrant (Ph 1b)
  Interventions: Drug: Abemaciclib
- Capivasertib Plus Fulvestrant and Investigator's choice of CDK4/6i (palbociclib or ribociclib) (Experimental): Capivasertib Plus Fulvestrant and Investigator's choice of CDK4/6i (palbociclib or ribociclib) (Ph III)
  Interventions: Drug: Capivasertib
- Fulvestrant and Investigator's choice of CDK4/6i (palbociclib or ribociclib) (Active Comparator): Fulvestrant and investigator's choice of CDK4/6i (palbociclib or ribociclib) (Ph III)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Capivasertib — Phase Ib: Capivasertib 320 mg/ 400 mg administered PO BD 4 days on /3 days off per week for 4 weeks (28 days cycle) Phase III: : Capivasertib, administered PO BD 4 days on / 3 days off per week for 4 weeks (28 days cycle) at the dose confirmed in the phase Ib portion
  Arms: Capivasertib Plus Fulvestrant and Investigator's choice of CDK4/6i (palbociclib or ribociclib); Capivasertib Plus Palbociclib and Fulvestrant
Drug: Fulvestrant — Phase Ib and Phase III: 500 mg (2 injections of 250 mg) on Day 1 of Weeks 1 and 3 of Cycle 1, and then on Day 1, Week 1 of each cycle thereafter
  Arms: Capivasertib Plus Palbociclib and Fulvestrant; Fulvestrant and Investigator's choice of CDK4/6i (palbociclib or ribociclib)
Drug: Palbociclib — Phase Ib: 100 mg/ 125 mg. Once daily for 21 consecutive days followed by 7 days off treatment to comprise a complete 28-day cycle Phase III: Administered once daily for 21 days of 28-day cycle, at the dose of 125 mg.
  Arms: Capivasertib Plus Palbociclib and Fulvestrant
Drug: Ribociclib — Phase Ib: 200 mg/ 400 mg/ 600 mg. Once daily for 21 consecutive days followed by 7 days off treatment to comprise a complete 28-day cycle Phase III: Administered once daily for 21 days of 28-day cycle, at the dose confirmed in the phase 1b portion.
  Arms: Capivasertib Plus Ribociclib and Fulvestrant
Drug: Abemaciclib — Phase Ib: 50 mg/ 100 mg/ 150 mg. Twice daily for 28 consecutive days to comprise a complete 28-day cycle
  Arms: Capivasertib Plus Abemaciclib and Fulvestrant

SUMMARY:
A Phase Ib/III Open-label, Randomised Study of Capivasertib plus CDK4/6 Inhibitors and Fulvestrant versus CDK4/6 Inhibitors and Fulvestrant in Hormone Receptor-Positive and Human Epidermal Growth Factor Receptor 2-Negative Locally Advanced, Unresectable or Metastatic Breast Cancer (CAPItello-292)

DETAILED DESCRIPTION:
This Phase Ib/III study (CAPItello-292) aims to evaluate the efficacy, safety and the degree of added benefit of capivasertib combined with CDK4/6i and fulvestrant in participants with locally advanced (inoperable) or metastatic HR+/HER2- breast cancer. Although the dosing regimens of capivasertib + fulvestrant and of CDK4/6i + fulvestrant are established separately, the dose and schedule for the triplet combinations (capivasertib + CDK4/6i + fulvestrant) need to be confirmed. Therefore, the initial dose finding Phase Ib part of the study will determine the recommended Phase III doses (RP3D) of the triplet combinations. The Phase III part of the study will evaluate the efficacy, safety and the degree of added benefit of the triplet combinations of capivasertib and fulvestrant with investigator's choice of CDK4/6i (either palbociclib or ribociclib at safe and tolerable doses, once identified) in comparison with a control arm (fulvestrant + investigator's choice of CDK4/6i [palbociclib or ribociclib]) in a ER+ HER2- maC high risk population that did not receive prior endocrine therapy in the advanced setting.

ELIGIBILITY:
Key inclusion criteria for both phases:

1. Adult females (pre-/peri-/ and post-menopausal), and adult males.
2. Histologically confirmed HR+/ HER2- breast cancer determined from the most recent tumour sample (primary or metastatic) per the American Society of Clinical Oncology and College of American Pathologists guideline. To fulfil the requirement of HR+ disease, a breast cancer must express ER with or without co-expression of progesterone receptor.
3. Eligible for fulvestrant therapy and at least one of the following: palbociclib, ribociclib, or abemaciclib, as per local investigator assessment. Previous tolerance to specific CDK4/6 inhibitors and dose levels required.
4. Adequate organ and bone marrow functions.
5. Consent to provide a mandatory FFPE tumour sample.

Key inclusion criteria only for phase III:

1. Previous treatment with an ET (tamoxifen, AI, or oral SERD) as a single agent or in combination, with radiological evidence of breast cancer recurrence or progression while on, or within 12 months of, completing a (neo)adjuvant ET regimen.
2. Provision of mandatory blood samples at screening for central testing using an investigational ctDNA test to be stratified based on PIK3CA/AKT1/PTEN status.
3. Be eligible for fulvestrant and at least one out of palbociclib or ribociclib (depending on the available CDK4/6i options at time of enrolment), as per local investigator assessment.
4. Have measurable lesion(s) according to Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST v1.1) or, in the absence of measurable disease, lytic or mixed bone lesions that can be assessed by computed tomography (CT) or magnetic resonance imaging (MRI).

Key exclusion criteria for both phases:

1. History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence.
2. Radiotherapy within 2 weeks prior to study treatment initiation.
3. Major surgery or significant traumatic injury within 4 weeks of the first dose of study treatment.
4. Persistent toxicities (CTCAE Grade >1) caused by previous anticancer therapy, excluding alopecia. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention may be included (eg, hearing loss or peripheral sensory neuropathy) after consultation with the AstraZeneca study physician.
5. Spinal cord compression, brain metastases or leptomeningeal metastases unless these lesions are definitively treated (eg. radiotherapy, surgery) and clinically stable off steroids for management of symptoms for at least 4 weeks prior to study treatment initiation.
6. Any of the following cardiac criteria at screening:

   (a). Mean resting corrected QT interval (QTcF): (i) Participants to be treated with palbociclib:: QTcF ≥ 470 ms obtained from the average of 3 consecutive (triplicate) ECGs (ii) Participants to be treated with ribociclib: QTcF ≥ 450 ms obtained from the average of 3 consecutive (triplicate) ECGs (iii) Participants to be treated with abemaciclib (Phase Ib only): QTcF ≥ 470 ms obtained from the average of 3 consecutive (triplicate) ECGs (b). Any clinically important abnormalities in cardiac rhythm, conduction or morphology of resting ECG (eg, complete left bundle branch block, third-degree heart block) (c). Any factors that increase the risk of QTc prolongation or risk of arrhythmic events (d). Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, unstable angina pectoris, congestive heart failure New York Heart Association (NYHA) grade ≥ 2 (e). Uncontrolled hypotension (f) uncontrolled hypertension (g). Cardiac ejection fraction outside institutional range of normal or < 50% (whichever is higher)
7. uncontrolled or high grade or symptomatic arrhythmia and atrial fibrillation
8. Any of these clinically significant abnormalities of glucose metabolism at screening:

   1. . diabetes mellitus type I or type II requiring insulin treatment
   2. . Glycated haemoglobin (HbA1c) ≥ 8.0% (63.9 mmol/mol)
9. Previous allogeneic bone marrow transplant or solid organ transplant.

Key exclusion criteria for the phase III only:

1. Any prior treatment with, AKT, PI3K or mTOR inhibitors.
2. Prior treatment with CDK4/6 inhibitors in the metastatic setting (prior CDK4/6 inhibitors permitted in the adjuvant setting provided there was a CDK4/6i treatment free interval of at least 12 months).
3. More than 1 line of chemotherapy for metastatic disease.
4. Any line of endocrine-based therapy for inoperable locally advanced or metastatic disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 895 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-08-14 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: 1. The number of participants with dose-limiting toxicity, as defined in the protocol. | Within the first 28 day cycle.
  Dose-limiting toxicity as described in the protocol that is not related to disease progression, intercurrent illness or concomitant medications and that, despite optimal therapeutic intervention, meets protocol-defined criteria.
Phase Ib: 2. The number of participants with treatment-related adverse events. | From baseline up to approximately 36 months.
  Data will include clinical observations, ECG parameters, clinical chemistry and haematology and vital signs assessed as the number of participants with treatment-related adverse events.
Phase Ib: 3. The number of participants with treatment-related serious adverse events. | From baseline up to approximately 36 months.
  Data will include clinical observations, ECG parameters, clinical chemistry and haematology and vital signs assessed as the number of participants with treatment-related adverse events.
Phase III: 1. Progression Free Survival (PFS). | Up to approximately 47 months.
  Progression Free Survival (PFS) is defined as time from randomization until progression per RECIST v1.1. as assessed by BICR or death due to any cause in the overall population, the altered population, and the confirmed non-altered population. RECIST related endpoints such as PFS, ORR, DoR, CBR will be collected.

SECONDARY OUTCOMES:
Phase Ib: 1. PK parameters for Palbociclib, Ribociclib, Abemaciclib: Cmax. | Cycle 0 (Cycle 0 is 3 days), Cycle 1 Day 11 and Cycle 1 Day 14 (Cycle 1 is 28 days).
  Maximum observed plasma (peak) drug concentration.
Phase Ib: 2. PK parameters for Palbociclib, Ribociclib, Abemaciclib: AUC0-72h. | Cycle 0 (Cycle 0 is 3 days).
  Partial area under the plasma concentration-time curve from zero to 72 hours post-dose.
Phase Ib: 3. PK parameters for Palbociclib, Ribociclib, Abemaciclib: AUC0-24h. | Cycle 0 (Cycle 0 is 3 days), Cycle 1 Day 11 and Cycle 1 Day 14 (Cycle 1 is 28 days).
  Partial area under the plasma concentration-time curve from zero to 24 hours post-dose.
Phase Ib: 4. PK parameters for Palbociclib, Ribociclib, Abemaciclib: Cmin. | Cycle 1 Day 11 and Cycle 1 Day 14 (Cycle 0 is 3 days and Cycle 1 is 28 days).
  Minimum observed plasma drug concentration.
Phase Ib: 5. PK parameters for capivasertib: Cmax. | Cycle 1 Day 11 (Cycle 0 is 3 days and Cycle 1 is 28 days).
  Maximum observed plasma (peak) drug concentration.
Phase Ib: 6. PK parameters for capivasertib: AUC0-12h. | Cycle 1 Day 11 (Cycle 0 is 3 days and Cycle 1 is 28 days).
  Partial area under the plasma concentration-time curve from zero to 12 hours post-dose.
Phase Ib: 7. PK parameters for capivasertib: Cmin. | Cycle 1 Day 11 (Cycle 0 is 3 days and Cycle 1 is 28 days).
  Minimum observed plasma drug concentration.
Phase Ib: 8. Objective Response Rate (ORR). | Up to approximately 36 months.
  Objective Response Rate (ORR) is defined as the proportion of patients with measurable disease at baseline who have a confirmed complete response (CR) or confirmed partial response (PR), as determined by the investigator at local site per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Phase Ib: 9. Clinical Benefit Rate (CBR) at 24 weeks. | Up to approximately 36 months.
  Clinical Benefit Rate (CBR) 24 weeks is defined as the percentage of patients who have a CR or PR or who have SD per RECIST v1.1 as assessed by the investigator at local site for at least 23 weeks after date of first dose.
Phase Ib: 10. Duration of Response (DoR). | Up to approximately 36 months.
  Duration of Response (DoR) will be defined as the time from the date of first documented confirmed response until date of documented progression per RECIST v1.1 as assessed by the investigator at local site or death due to any cause.
Phase Ib: 11. Progression Free Survival (PFS). | Up to approximately 36 months.
  Progression Free Survival (PFS) is defined as time from date of first dose until progression per RECIST v1.1. as assessed by the investigator at local site or death due to any cause.
Phase III: 1. Overall Survival (OS). | Up to approximately 69 months.
  Overall survival (OS) - time from randomization until the date of death due to any cause, secondary outcome measure in participants with HR+/HER2- locally advanced or metastatic breast cancer with gene alteration in PIK3CA/AKT1/PTEN - altered population, confirmed non-altered population and overall population.
Phase III: 2. Objective Response Rate (ORR). | Up to approximately 47 months.
  Objective Response Rate (ORR) - the proportion of patients who have a complete or partial response, as determined by BICR per RECIST v1.1 in participants with HR+/HER2- locally advanced or metastatic breast cancer with gene alteration in PIK3CA/AKT1/PTEN - altered population, confirmed non-altered population and overall population.
Phase III: 3. Progression Free Survival 2 (PFS2) | Up to approximately 69 months.
  Progression Free Survival 2 (PFS2) - time from randomization to the earliest of the progression event, after first subsequent therapy or death.
Phase III: 4. Duration of Response (DoR). | Up to approximately 47 months.
  Duration of Response (DoR) - the time from the date of first documented response until the date of progression per RECIST v1.1 as assessed by BICR, or death due to any cause.
Phase III: 5. Clinical Benefit Rate (CBR) at 24 weeks. | Up to approximately 47 months.
  Clinical Benefit Rate (CBR) at 24 weeks-the % of patients who have a CR or PR or who have SD per RECIST v1.1 as assessed by BICR for at least 23 weeks after randomisation.
Phase III: 6. Participant-reported physical functioning | Up to approximately 69 months.
  TTD of physical functioning as measured by the physical functioning subscale of the EORTC QLQ-C30.
Phase III: 7. Participant-reported GHS/QoL in participants | Up to approximately 69 months.
  TTD of GHS/QoL as measured by the GHS/QoL subscale of the EORTC QLQ-C30.
Phase III: 8. Participant-reported overall side effect bother in participants in the capivasertib arm relative to control arm | Up to approximately 69 months.
  Proportion of participants experiencing different levels of overall treatment tolerability as measured by the Patient Global Impression-Treatment Tolerability (PGI-TT).
Phase III: 9. Plasma concentration of capivasertib pre- and post-dose. | Up to approximately 69 months.
  Plasma concentration of capivasertib pre-, and post-dose.
Phase III: 10. The number of participants with adverse events. | Up to approximately 69 months.
  Data will include clinical observations, ECG parameters, clinical chemistry / haematology / glucose metabolism parameters and vital signs assessed as the number of participants with adverse events.
Phase III: 11. The number of participants with serious adverse events. | Up to approximately 69 months.
  Data will include clinical observations, ECG parameters, clinical chemistry / haematology / glucose metabolism parameters and vital signs assessed as the number of participants with serious adverse events.

CONTACTS AND LOCATIONS:
Locations (239):
- United States (48):
  - Research Site, Tucson, Arizona
  - Research Site, Fountain Valley, California
  - Research Site, Glendale, California
  - Research Site, Los Angeles, California
  - Research Site, Napa, California
  - Research Site, Newport Beach, California
  - Research Site, San Francisco, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Rosa, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Quincy, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Hannibal, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Camden, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Gresham, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Greenville, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Falls Church, Virginia
  - Research Site, Leesburg, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Tacoma, Washington
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Chivilcoy
  - Research Site, Rosario
  - Research Site, Santa Fe
- Australia (5):
  - Research Site, Darlinghurst
  - Research Site, Miranda
  - Research Site, Nedlands
  - Research Site, Wahroonga
  - Research Site, Waratah
- Belgium (5):
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Haine-Saint-Paul
  - Research Site, Leuven
- Brazil (9):
  - Research Site, Alfenas
  - Research Site, Blumenau
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Porto Velho
  - Research Site, São Paulo
  - Research Site, Taubaté
  - Research Site, Teresina
  - Research Site, Vitória
- Canada (12):
  - Research Site, Abbotsford, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Sherbrooke, Quebec
  - Research Site, Chicoutimi
  - Research Site, Montreal
- China (22):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiangyang
  - Research Site, Xuzhou
  - Research Site, Zhengzhou
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Hillerød
  - Research Site, Odense
- France (8):
  - Research Site, Bobigny
  - Research Site, Clermont-Ferrand
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Plérin
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- Germany (21):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Bottrop
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Georgsmarienhütte
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heilbronn
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Mannheim
  - Research Site, Mönchengladbach
  - Research Site, Münster
  - Research Site, Regensburg
  - Research Site, Stade
  - Research Site, Trier
  - Research Site, Ulm
- India (9):
  - Research Site, Bangalore
  - Research Site, Jaipur
  - Research Site, Mohali
  - Research Site, Mysuru
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Puducherry
  - Research Site, Vadodara
  - Research Site, Varanasi
- Italy (12):
  - Research Site, Aviano
  - Research Site, Bologna
  - Research Site, Catanzaro
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Misterbianco
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Prato
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (24):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Isehara-shi
  - Research Site, Kagoshima
  - Research Site, Kōtoku
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Naha
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shimotsuke-shi
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Takasaki-shi
  - Research Site, Tsu
  - Research Site, Yokohama
- Malaysia (5):
  - Research Site, George Town
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
  - Research Site, Pulau Pinang
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Rzeszów
  - Research Site, Warsaw
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Santiago de Compostela
- Sweden (3):
  - Research Site, Lund
  - Research Site, Solna
  - Research Site, Vaxjo
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Dusit
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Lampang
  - Research Site, Ratchathewi
- Turkey (Türkiye) (7):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Goztepe Istanbul
  - Research Site, Karşıyaka
  - Research Site, Kayseri
  - Research Site, Malatya
  - Research Site, Samsun
- United Kingdom (5):
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Londonderry
  - Research Site, Taunton
  - Research Site, York
- Vietnam (5):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hồ Chí Minh
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Breast Cancer Study Locator details (for US) — https://www.breastcancerstudylocator.com/trial/listing/284051